CLINICAL TRIAL: NCT01513005
Title: Feasibility of Day Case Management by Laparoscopic Sleeve Gastrectomy for Obesity: a Pilot Study
Brief Title: Feasibility of Laparoscopic Sleeve Gastrectomy in Day Case Surgery
Acronym: GASTRAMBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI10-PR.-REGIMBEAU; 2010-A01178-31 (Other: ID-RCB)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Laparoscopic Sleeve Gastrectomy; obesity management
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laparoscopic Sleeve Gastrectomy (Experimental)
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Sleeve Gastrectomy — the operative technique consists in few steps:
  * position of 4 trocars and insertion of a nasogastric tube
  * dissection and mobilization of the greater curvature of the stomach
  * preparation of the stomach for division
  * gastric partition
  * extraction of the gastric remnant
  * postoperative surveillance

SUMMARY:
The aim of this study is to determinate the feasibility of the Laparoscopic Sleeve Gastrectomy, a bariatric surgery i.e. a surgery as a treatment for obesity, could be proposed as a Day-Case surgery.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether the patients with morbid obesity requiring a surgical approach by Laparoscopic Sleeve Gastrectomy could be operated according to a "day-case surgery" modality.

The sequence of this study is the following:

1. patients consultation for bariatric management: during this consultation, the investigator is looking for exclusion criteria and prescribes laboratory tests.
2. medical records of each patient are reviewed by an obesity-related staff: Laparoscopic Sleeve Gastrectomy is proposed.
3. during a second consultation, the surgeon informed the patient about the proposition of the staff and his potential inclusion in this study
4. after obtained his consent, the surgical procedure is planned and Laparoscopic Sleeve Gastrectomy is done in the Day-Case Surgery Unit.
5. the following day the surgery, a nurse calls the patient to identify a potential postoperative outcome (nausea, vomiting, uncontrolled pain...)
6. the 8th postoperative day, a consultation is done with laboratory tests and dietary follow-up.
7. follow-up consultations are scheduled at 3, 6 and 12 months to evaluate the efficiency of the surgery procedure.

ELIGIBILITY:
Inclusion Criteria:

* sufficient understanding
* good observance of medical prescription
* availability of a responsible adult for the first operative night
* patients living nearby the hospital (1 h maximum away)
* telephonic accessibility
* between 18 and 60 years old adults
* body mass index less than 60 kg/m2
* obesity requiring bariatric surgery
* surgery validated by an obesity-related staff

Exclusion Criteria:

* patient under administrative or legal protection
* obesity without HAS criteria
* cardiovascular comorbidity
* pulmonary comorbidity
* curative anticoagulant therapy
* bad diabetes control
* body mass index higher than 60 kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
unexpected admission rate | the day following the surgery
  the unexpected admission rate corresponds to the number of overnight hospitalization i.e. the number of patients not treated considering a Day-Case Surgery.

SECONDARY OUTCOMES:
readmission rate | one year
  the readmission rate is defined as the number of readmission with conventional hospitalization
unexpected consultation rate | one year
  the unexpected consultation rate corresponds to the number of consultations after the Laparoscopic Sleeve Gastrectomy because of a postoperative outcome (adverse event, pain...)
reoperation rate | one year
overall length of stay | one year
  the overall length of stay corresponds to the duration of all hospitalizations i.e. between the surgical procedure and the end of follow up.
per operative outcomes | one year
  the per operative outcomes include each event observed during the surgical procedure
postoperative outcomes | one year
  the postoperative outcomes include all outcomes reported during the follow-up period
efficiency of Laparoscopic Sleeve Gastrectomy | six months
  the efficiency of Laparoscopic Sleeve Gastrectomy is evaluated with the BAROS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc REGIMBEAU, MD,phD, Principal Investigator — CHU Amiens
Locations (1):
- North Universitary Hospital, Amiens, France

REFERENCES:
- [Background] Pequignot A, Dhahria A, Mensah E, Verhaeghe P, Badaoui R, Sabbagh C, Regimbeau JM. Stapling and Section of the Nasogastric Tube during Sleeve Gastrectomy: How to Prevent and Recover? Case Rep Gastroenterol. 2011;5(2):350-4. doi: 10.1159/000329706. Epub 2011 Jul 6. PMID 21769286
- [Background] Dhahri A, Verhaeghe P, Hajji H, Fuks D, Badaoui R, Deguines JB, Regimbeau JM. Sleeve gastrectomy: technique and results. J Visc Surg. 2010 Oct;147(5 Suppl):e39-46. doi: 10.1016/j.jviscsurg.2010.08.016. No abstract available. PMID 20971049
- [Background] Sabbagh C, Verhaeghe P, Dhahri A, Brehant O, Fuks D, Badaoui R, Regimbeau JM. Two-year results on morbidity, weight loss and quality of life of sleeve gastrectomy as first procedure, sleeve gastrectomy after failure of gastric banding and gastric banding. Obes Surg. 2010 Jun;20(6):679-84. doi: 10.1007/s11695-009-0007-4. Epub 2009 Nov 10. PMID 19902316
- [Background] Fuks D, Verhaeghe P, Brehant O, Sabbagh C, Dumont F, Riboulot M, Delcenserie R, Regimbeau JM. Results of laparoscopic sleeve gastrectomy: a prospective study in 135 patients with morbid obesity. Surgery. 2009 Jan;145(1):106-13. doi: 10.1016/j.surg.2008.07.013. Epub 2008 Sep 30. PMID 19081482
- [Background] Fuks D, Dumont F, Berna P, Verhaeghe P, Sinna R, Sabbagh C, Demuynck F, Yzet T, Delcenserie R, Bartoli E, Regimbeau JM. Case report-complex management of a postoperative bronchogastric fistula after laparoscopic sleeve gastrectomy. Obes Surg. 2009 Feb;19(2):261-264. doi: 10.1007/s11695-008-9643-3. Epub 2008 Aug 12. PMID 18696169
- [Result] Badaoui R, Alami Chentoufi Y, Hchikat A, Rebibo L, Popov I, Dhahri A, Antoun G, Regimbeau JM, Lorne E, Dupont H. Outpatient laparoscopic sleeve gastrectomy: first 100 cases. J Clin Anesth. 2016 Nov;34:85-90. doi: 10.1016/j.jclinane.2016.03.026. Epub 2016 May 3. PMID 27687352